CLINICAL TRIAL: NCT03520829
Title: Protocol for Evaluating a Planning Algorithm for Gamma Knife Radiosurgery
Acronym: SPEED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-52; 2017-A02753-50 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-04-27; First posted 2018-05-11 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Vestibular Schwannoma; Brain Metastases; Para-optic Meningioma
MeSH Terms: conditions — Neuroma, Acoustic; Brain Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient treated for Gamma Knife
  Interventions: Device: Intuitive Plan

INTERVENTIONS:
Device: Intuitive Plan — dosimetric planning software

SUMMARY:
The process of developing Gamma Knife radiosurgery treatment plans is today very dependent on the level of human expertise resulting in a great heterogeneity of the intrinsic qualities of the treatment planning and the quality of care delivered in radiosurgery.

The existing reverse planning systems, although they have progressed considerably in recent years, produce results that are still lower than those achieved by an expert.

Conventionally, an experienced dosimetric planner will act mainly on the coordinates of the position of the isocenters, on the size of the collimators, sector by sector, and on the irradiation time of each isocenters. In theory, the combination of these variables provides access to billions of combinatorics whose diversity far exceeds the computational capabilities of the human mind. The dosimetric planner therefore uses a very small part of the spectrum of possible patterns by always reproducing a limited number of empirical solutions.

The company Intuitive Therapeutics has developed a new mathematical algorithm which can automatically test in a very short time all the combinatorial possibilities and converge very quickly to the solution that best meets the clinical, anatomical and dosimetric objectives defined by the neurosurgeon. The quick processing of the system also allows the operator to modify the constraints to refine the proposed result in real time.

The demonstration of the reality of the performances of this algorithm would give the ability to even inexperienced users to develop high performance planning for the benefit of the patient in terms of optimizing the efficacy / toxicity ratio of the radiosurgery treatment results

The primary objective is to evaluate comparatively the quality of the schedules produced by the algorithm developed by the company Innovative Therapeutics to those produced by an expert who carried out more than 15000 dosimetric plannings and radiosurgical interventions.

The main criterion of comparison is the Paddick index.

The secondary criteria for comparison are:

* Compliance index
* selectivity index
* Gradient index
* Maximum, minimum, average dose at risk structures
* Dose distribution in the target volume
* Treatment time (at equal source activity)
* Time of realization of the planning

It was chosen to treat patients with vestibular Schwannoma OR multiple brain metastases (> 5) treated in single session by Gamma Knife OR para-optic meningioma in hypo-fractionated treatment on Gamma Knife with restraint mask with inclusion of visual paths in the target volume planning.

The aim of the study is to show at least the non-inferiority of this new method compared to the expert user based on the Paddick Index. This index has continuous values between 0 and 1, 0 being the worst case and 1 being the ideal solution. In order to define the sample size needed for each pathology, a pilot phase is required. This phase can be performed retrospectively using treatments already defined by the expert user. This pilot phase will allow us to identify the difference that can be expected between the index values and the variability of this difference. Based on these values we will be able to determine the size of the sample allowing us to statistically test the non-inferiority, or even the superiority of this new device. The number of cases to be included during the pilot phase should be at least ten cases and a maximum of thirty cases. The choice of the number of cases to be integrated during this pilot phase will depend on the homogeneity of the differences obtained on the first cases. These values will allow us to calculate the size of the samples necessary for the study of non-inferiority as well as for the study of superiority. Depending on the calculated sizes samples we will make a choice to ensure that this study takes place in the expected duration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old
* Patient treated for Gamma Knife
* Patient who has benefited or needs Gamma-Knife radiosurgical treatment
* Patient affiliated to a social protection scheme.
* Patient having understood the information notice and expressed his non opposition.

Exclusion Criteria:

* Patient with a contraindication to perform a brain MRI
* Patient with a contraindication to radiosurgical treatment (previous treatment with cerebral radiotherapy)
* Pregnant and lactating women
* Simultaneous participation in another therapeutic trial or in the exclusion period of a previous clinical trial.
* Vulnerable persons: minors, protected adults (guardianship or trusteeship) and adults unable to express their consent.
* Patient expressing opposition to participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single-session treated patient with vestibular schwannoma or multiple brain metastases (> 5) or para-optic meningioma
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-01-10 (Estimated); Study Completion 2020-01-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate comparatively the quality of the schedules produced by the algorithm developed | one year
  to show at least the non-inferiority of this new method compared to the expert user based on the Paddick Index. This index has continuous values between 0 and 1, 0 being the worst case and 1 being the ideal solution

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — ASSISTANCE PUBLIQUE HÔPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No